CLINICAL TRIAL: NCT06946628
Title: Combination Therapy With Semaglutide, Empagliflozin and Pioglitazone Versus Standard Therapy in Newly Diagnosed Type 2 Diabetes: a Multi-center Randomized Controlled Trial
Brief Title: New Triple Therapy in Newly Diagnosed Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, Director of Endocrinology Department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: New Triple-2025
Record Dates: First submitted 2025-03-03; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Group A (triple combination therapy group): semaglutide, empagliflozin, and pioglitazone treatment.
  Group B (standard therapy group): metformin-based treatment is recommended when not contraindicated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (triple combination therapy group) (Experimental): semaglutide, empagliflozin, and pioglitazone treatment. 1) Initiate with Semaglutide 0.25 mg once weekly (qw) + Empagliflozin 10 mg once daily (qd) + Pioglitazone 15 mg once daily (qd); 2) After 1 month, if blood glucose is not controlled, adjust to Semaglutide 0.5 mg qw + Empagliflozin 20 mg qd + Pioglitazone 30 mg qd. If Semaglutide is well-tolerated, increase to 1 mg qw after 1 week; 3)If blood glucose remains uncontrolled after 1 month, add basal insulin therapy.
  Interventions: Drug: Group A (triple combination therapy group)
- Group B (standard therapy group) (Active Comparator): metformin-based treatment is recommended when not contraindicated. 1).Initiate with Metformin monotherapy, titrate to the target dose of 1000 mg twice daily (bid) within 1 month or to the maximum tolerated dose (if Metformin is not tolerated, switch to Linagliptin 5 mg qd); 2) After 1 month, if blood glucose is not controlled, add a second antidiabetic drug, Empagliflozin 20 mg qd; 3) After another month, if blood glucose remains uncontrolled, add Semaglutide 0.25 mg qw, then increase to 0.5 mg qw after 1 month. If well-tolerated, increase to 1.0 mg qw after 1 week; 4) If blood glucose remains uncontrolled after 1 month, add basal insulin therapy.
  Interventions: Drug: Group B (standard therapy group)

INTERVENTIONS:
Drug: Group A (triple combination therapy group) — 1) Initiate with Semaglutide 0.25 mg once weekly (qw) + Empagliflozin 10 mg once daily (qd) + Pioglitazone 15 mg once daily (qd); 2) After 1 month, if blood glucose is not controlled, adjust to Semaglutide 0.5 mg qw + Empagliflozin 20 mg qd + Pioglitazone 30 mg qd. If Semaglutide is well-tolerated, increase to 1 mg qw after 1 week; 3)If blood glucose remains uncontrolled after 1 month, add basal insulin therapy.
  Arms: Group A (triple combination therapy group)
Drug: Group B (standard therapy group) — metformin-based treatment is recommended when not contraindicated. 1).Initiate with Metformin monotherapy, titrate to the target dose of 1000 mg twice daily (bid) within 1 month or to the maximum tolerated dose (if Metformin is not tolerated, switch to Linagliptin 5 mg qd); 2) After 1 month, if blood glucose is not controlled, add a second antidiabetic drug, Empagliflozin 20 mg qd; 3) After another month, if blood glucose remains uncontrolled, add Semaglutide 0.25 mg qw, then increase to 0.5 mg qw after 1 month. If well-tolerated, increase to 1.0 mg qw after 1 week; 4) If blood glucose remains uncontrolled after 1 month, add basal insulin therapy.
  Arms: Group B (standard therapy group)

SUMMARY:
The goal of this clinical trial is to learn the efficany of combination therapy with semaglutide, empagliflozin and pioglitazone versus standard therapy in newly diagnosed type 2 diabetes. The main objectives to achieve are:

1. To compare efficacy of the triple combination therapy against standard therapy in achieving type 2 diabetes remission in patients newly diagnosed with T2DM.
2. To compare the effects on β-cell function and glycemic control of the triple combination therapy against standard therapy in patients newly diagnosed with T2DM

Researchers will compare drug new triple combination therapy with semaglutide, empagliflozin, and pioglitazone to standard therapy (metformin-based treatment) to see if new triple combination therapy works better in achieving type 2 diabetes remission .

Participants will:

1. Take new triple combination therapy or a standard therapy every day for 6 months
2. Visit the clinic once every 0.5-1 month for checkups and tests
3. Keep a diary of their fingertip blood glucose and adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years≤age≤75 years at the time of signing informed consent.
2. Newly diagnosed with type 2 diabetes, or diagnosed within 1 years according to the WHO diagnostic criteria.
3. Individuals who had not received previous antidiabetic therapy, or had not received antidiabetic therapy within 3 months prior to screening, or had not received antidiabetic therapy for more than 3 consecutive months or a combined total of more than 3 months in the past 2 years.
4. 6.5%≤HbA1c≤9.0% at screening confirmed by central laboratory analysis.
5. BMI≥24 kg/m2.

Exclusion Criteria:

1. Individuals with type 1 diabetes or special types of diabetes.
2. Allergy or intolerance to investigational drugs.
3. Estimated Glomerular Filtration Rate (eGFR) <20 mL/min/1.73 m².
4. Individuals with heart failure in New York Heart Association [NYHA] class III or IV in the 6 months prior to randomization.
5. History of bladder cancer or hematuria.
6. History of Multiple Endocrine Neoplasia Type 2 (MEN 2) or relevant family history.
7. History or family history of Medullary Thyroid Carcinoma (MTC), or susceptibility to MTC due to hereditary conditions.
8. History of fasting blood glucose≥13.9 mmol/L or the necessity for insulin use due to severe infection, diabetic foot, etc.
9. History of acute diabetic complications: including diabetic ketoacidosis, hyperglycemic hyperosmolar state, lactic acidosis.
10. Severe diabetic microvascular complications: proliferative retinopathy, or urinary AER>300mg/g, or urinary protein positive, quantitative >0.5g/24h.
11. Uncontrolled painful diabetic neuropathy and significant diabetic autonomic neuropathy.
12. Severe diabetic macrovascular complications: myocardial infarction, stroke or hospitalization for unstable angina and/or transient ischemic attack and/or peripheral arterial disease required for vascular intervention or amputation within the 12 months prior to screening.
13. Blood pressure persistently higher than 180/110 mmHg and not controllable to ≤160/100 mmHg within 1 week.
14. Alanine Aminotransferase (ALT) ≥2.5 times the upper normal limit, total bilirubin ≥1.5 times the upper normal limit.
15. Hemoglobin <100g/L or requiring regular blood transfusion.
16. Use of medicines potentially affecting blood glucose for more than 1 week cumulatively in the past 12 weeks, such as corticosteroids, growth hormone analogs, estrogen/progestogen, high-dose diuretics, antipsychotic drugs, etc.
17. Participation in another trial involving medicine therapy within the past 3 months.
18. Expected lifespan less than 2 years as per the investigator's clinical judgment, e.g., but not limited to malignancy.
19. Pregnant or lactating females, or females of childbearing potential who cannot or are unwilling to use adequate contraception.
20. Deemed unsuitable for participation in this clinical trial at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetic remission rate | 6 months after discontinuation of medication
  Diabetic remission rate at 6 months after discontinuation of medication (percentage of patients with HbA1c <6.5% at 6 months after discontinuation of medication)

SECONDARY OUTCOMES:
Diabetic remission rate | 3 and 12 months after discontinuation of medication
  Diabetic remission rate at 3 and 12 months after discontinuation of medication and the time of diabetic remission
Time required to achieve glycemic goal | 6 months of medication
  The time required to achieve glycemic goal(FBG <6.1mmol/L, 2h PPG <8.0mmol/L or HbA1c<6.5%)
EQ-5D-5L questionnaires, quality of life | At baseline, at 6 months of medication treatment, and at 3, 6, and 12 months after discontinuation of medication
  EQ-5D-5L questionnaires, assessment of quality of life. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Incremental cost per additional remission | 6 months after discontinuation of medication
  Incremental cost per additional remission at 6 months after discontinuation of medication
HbA1c | baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
  HbA1c level at baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
Blood glucose level | baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
  Fasting and 2-hour postprandial blood glucose level at baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
Blood insulin level | baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
  Fasting and 2-hour postprandial insulin level at baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
Blood C-peptide level | baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
  Fasting and 2-hour postprandial C-peptide level at baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
Pancreatic β-cell function | baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
  HOMA-B at baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
Insulin resistance | baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
  HOMA-IR at baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
Weight changes | baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
  Weight at baseline, at 6 months of medication, and at 3, 6, and 12 months after discontinuation of medication
Time in range (TIR) | At baseline, at 6 months of medication treatment, and at 6 months after discontinuation of medication
  Time within the target blood glucose range (3.9-10.0 mmol/L)
Incremental cost per additional improvement in Time in Range (TIR) | 6 months of medication treatment, and at 6 months after discontinuation of medication
  Incremental cost per additional improvement in Time in Range (TIR) at 6 months of medication treatment, and at 6 months after discontinuation of medication
Incremental cost per QALY gained | at baseline, at 6 months of medication treatment, and at 3, 6, and 12 months after discontinuation of medication
  Incremental cost per QALY gained, derived from EQ-5D-5L assessments at baseline, at 6 months of medication treatment, and at 3, 6, and 12 months after discontinuation of medication

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No